CLINICAL TRIAL: NCT03582878
Title: Effect of Sirolimus or Mycophenolate With Tacrolimus on Survival of Pancreas and Kidney Grafts in Type 1 Diabetic Recipients After Simultaneous Pancreas and Kidney Transplantation
Brief Title: Sirolimus vs Mycophenolate With Tacrolimus in Simultaneous Pancreas and Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Frantisek Saudek, professor, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SiroMMFStudy 1
Record Dates: First submitted 2018-04-25; First posted 2018-07-11 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mycophenolate mofetil (Active Comparator): mycophenolate mofetil dosing 1g before transplantation and 1g bid afterwards
  Interventions: Drug: Mycophenolate Mofetil
- Sirolimus (Experimental): Sirolimus oral product Dosing 5mg orally 2-6h before transplantation Target trough levels between 5-10ng/ml
  Interventions: Drug: Sirolimus Oral Product

INTERVENTIONS:
Drug: Sirolimus Oral Product — Oral form of sirolimus, daily dosing to achieve target trough levels between 5-10ng/ml since 1.day of transplantation
  Other Names: Rapamune
  Arms: Sirolimus
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil dosing 1g before transplantation and 1g bid afterwards
  Other Names: CellCept
  Arms: mycophenolate mofetil

SUMMARY:
This is prospective randomized open single center clinical study to compare effect of sirolimus vs mycophenolate tacrolimus based protocol on pancreas and kidney graft survival in simultaneous pancreas and kidney recipients.

DETAILED DESCRIPTION:
MTOR (mammalian target of rapamycin) inhibitors represent group of immunosuppressive drugs with mechanism of T-cell blockade complementary to calcineurin inhibitors. The investigators presume that combination of sirolimus with tacrolimus will result in better survival of pancreatic and kidney grafts in simultaneous pancreas and kidney transplantations.

The study is proposed as a single-center extension of EUROSPK 002 trial originally started in 2004 by the EUROSPK Study Group. Recruitment of recipients started in 2004 with approval of EUROSPK 002. The patient recruitment has continued in a single center (Institute for Clinical and Experimental Medicine in Prague, Czech Republic) using the same inclusion and exclusion criteria. The recipients of primary kidney and pancreas transplantation have been randomized into 2 arms.

* In the intervention arm sirolimus is added to protocol at a dose of 5 mg immediately before transplantation, the dose is adjusted to maintained trough sirolimus trough levels between 5-10ng/ml.
* In the control arm mycophenolate mofetil was added to tacrolimus. Starting with 1g before transplantation, the dose has been increased to 1g bid afterwards.

Induction protocol at day 0. consists of ATG (antithymocyte globulin)induction 8mg/kg , Tacrolimus 0.05mg/kg, Methylprednisolone 125mg. Dosing of tacrolimus has been adjusted to maintain trough levels between 5-10ng/ml. ATG was administered at 3mg/kg on days 1.-3. Steroids have been gradually tapered from a dose of 20 mg prednison orally and withdrawn by 6w after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* End stage kidney failure
* Negative CDC crossmatch
* Female patients of childbearing age must have a negative pregnancy test
* Patient must have signed the Patient Informed Consent Form.
* Patient must receive a primary simultaneous pancreas/kidney (SPK) cadaver transplant,

Exclusion Criteria:

* Patient is pregnant or breastfeeding.
* Patient is allergic or intolerant to Mycophenolate Mofetil, Sirolimus, ATG, Tacrolimus
* Patient has malignancy or history of malignancy, with the exception of adequately treated localized squamous cell or basal cell carcinoma, without recurrence.
* Patient has been included in another clinical trial protocol for any investigational drug within 4 weeks prior to randomization.
* Patient has any form of substance abuse or psychiatric disorder or condition, which invalidate communication.
* Severe cardiac failure or severe liver failure diagnosed at the time of transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Pancreas graft survival | 10 years
  Number of failed pancreatic grafts, failure is defined as graft removal, death, retransplantation or return to intensified insulin regimen.

SECONDARY OUTCOMES:
Recipient survival | 10 years
  Long-term recipient survival evaluated with Kaplan-Meyer method
Wound healing time | 1year
  The number of days from transplantation to date of completely healed wound
Kidney graft survival | 10 years
  Number of failed kidneys evaluated with Kaplan-Meyer method. Failure defined as return to dialysis, death, retransplantation or graft removal

CONTACTS AND LOCATIONS:
Overall Officials: Frantisek Saudek, MD, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Girman P, Lipar K, Kocik M, Voska L, Koznarova R, Marada T, Lanska V, Saudek F. Sirolimus vs mycophenolate mofetil (MMF) in primary combined pancreas and kidney transplantation. Results of a long-term prospective randomized study. Am J Transplant. 2020 Mar;20(3):779-787. doi: 10.1111/ajt.15622. Epub 2019 Oct 23. PMID 31561278